CLINICAL TRIAL: NCT01780129
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group Multi-Center Phase II Clinical Study to Evaluate the Efficacy and Safety of HW6 in the Treatment of Traumatic/Hemorrhagic Shock and Septic Shock
Brief Title: Polydatin Injectable (HW6) for Shock Treatment
Acronym: PIST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neptunus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HW6-01-US; HW6-01-US (Registry Identifier: Neptunus Pharmaceuticals, Inc.)
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Shock, Hemorrhagic; Shock, Traumatic; Shock, Septic
MeSH Terms: conditions — Shock, Hemorrhagic; Shock, Traumatic; Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polydatin Injectable (HW6) (Experimental): 10ml(2 ampoules) diluted in 500ml of 0.9% NaCl solution for i.v. infusion over 2 hours; once daily for 5 consecutive days
  Interventions: Drug: Polydatin Injectable
- HW6 blank dummy (0.9%NaCl) (Placebo Comparator): 10ml (2 ampoules) diluted in 500ml of 0.9% NaCl solution for i.v. infusion over 2 hours; once daily for 5 consecutive days

INTERVENTIONS:
Drug: Polydatin Injectable — Dilute two 100mg/5mL vials of HW6 into 500mL 0.9% NaCl injection and administer as i.v. infusion over 2 hours. The drug should be given as early as possible right after the IC Form is signed on Day 1, and once every 24 hours for additional 4 doses.
  Other Names: HW6
  Arms: Polydatin Injectable (HW6)

SUMMARY:
HW6 can prolong animal's survival time and increase the survival rate. HW6 enhances cardiac function, improves microcirculation, and increases blood pressure and pulse pressure, and improves blood perfusion of important organs; HW6's anti-shock activity comes from a combined multiple target pharmacological effects.

Based on a completed phase II trial conducted in China, HW6 can effectively treatment shock patient.

This is a phase II clinical study to further evaluate the efficacy and safety of Polydatin Injectable 100mg/5mL/via (HW6) in the treatment of shock in the United States. Patients with traumatic/hemorrhagic shock or septic shock admitted to the emergency room or ICU with systolic blood pressure < 90mmHg, or is on vasopressor(s) for systolic blood pressure stabilization, regardless the types of completed, on-going, or projected Standard of Care or surgery will be recruited to participant in the trial. A total of 120 patients with traumatic/hemorrhagic shock and 120 patients with septic shock will be enrolled. For each type of shock, sixty patients each will be in test group and control group. Both adult males and females aged 18-80 years are eligible. The primary clinical endpoint is the time length (TL) between the start of HW6 administration to the onset of the first treatment success, that is: the systolic blood pressure is stabilized at ≥90mmHg and MAP≥65mmHg for 1 hour without the use of vasopressors. Several secondary endpoints and biomarkers will be measured.

Efficacy data will be compared using group t-test or Wilcoxon log-rank test between treatment groups and placebo groups. Safety data will also be reported accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females aged 18-80 years.
* Patients with traumatic/hemorrhagic shock or septic shock admitted to the emergency room or ICU with systolic blood pressure < 90mmHg, or is on vasopressor(s) for systolic blood pressure stabilization, regardless the types of completed, ongoing, or projected Standard of Care or surgery.
* Patients (or its relative) who have signed Informed Consent Form to voluntarily participate in this clinical study.

Exclusion Criteria:

* Has known allergic constitution or history of alcohol or drug allergy. or
* Complicating acute cardiac failure, acute renal failure, acute liver failure or disseminated intravascular coagulation (DIC). or
* Pregnant or lactating women. or
* Complicating moderate to severe craniocerebral injury. or
* Has known previous severe chronic disease(s) in liver, kidney, carvascualr system or central nervous system. or

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The time length (TL) between the start of HW6 administration to the onset of the first TS. | From the start of drug administration to the onset of TS (OTS) where the first systolic blood pressure≥90mmHg and MAP≥65mmHg is observed in the 7 consecutive measures
  Treatment success (TS): the systolic blood pressure is stabilized at ≥90mmHg and MAP≥65mmHg for 1 hour without the use of vasopressor(s).
  Blood pressure will be recorded every 10 min. Treatment success is considered to have been achieved when 7 consecutive systolic blood pressure to be≥90mmHg and MAP≥65mmHg.
  The TL is the time from the start of drug administration to the onset of TS (OTS) where the first systolic blood pressure≥90mmHg and MAP≥65mmHg is observed in the 7 consecutive measures.
  Blood pressure will be measured every hour after the TS. If blood pressure become unstable, standard care will be in practice.

SECONDARY OUTCOMES:
The amount and duration of total vasopressor(s) used during this TL period | From the start of drug administration to the onset of TS (OTS) where the first systolic blood pressure≥90mmHg and MAP≥65mmHg is observed in the 7 consecutive measures
  Observation period: From start of study drug treatment to OTS. Record the details of the use of vasopressor(s) during TL for each subject, including name of medication, infusion concentration and rate, and the duration of each concentration and rate being maintained.
  Duration of vasopressor(s) use: accurate to the minute, or by the cumulative time of each administration if used intermittently.
  Total dose of vasopressor(s)：The total dose of each vasopressor.
The degree of fluid dependence | from the start of testing drug to the OTS
Metabolic indicators | Within 6 days
  Arterial blood lactate, lactate clearance, oxygen saturation mixed venous blood, blood gas levels
Severity of organ dysfunction in the ICU | Daily during the administration stay after enrollment
  Compare the changes in SOFA score during the administration stay between the two groups to assess the protective effect of the study drug on vital organs.
Duration of ICU stay | The total time (in hours) of ICU admission from the day of administration to day 7 (7 days)
28-day survival | From the end of drug administration to Day 28

OTHER OUTCOMES:
Fluid intake and output volume | Every 24h for 5 days

CONTACTS AND LOCATIONS:
Overall Officials: YU Lin, PhD, Study Chair — Neptunus Pharmaceuticals Inc.
Locations (1):
- Christiana Care, Newark, Delaware, United States